CLINICAL TRIAL: NCT01242696
Title: PROMUS™ Element™ Everolimus-Eluting Coronary Stent System European Post- Approval Surveillance Study To Evaluate Real World Clinical Outcomes Data for the TAXUS® Element™ Coronary Stent System in Unselected Patients in Routine Clinical Practice
Brief Title: TAXUS® Element™ Paclitaxel-Eluting Coronary Stent System European Post-Approval Surveillance Study (TE-Prove)
Acronym: TE-Prove
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: S2059
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Heart Disease
Keywords: Drug Eluting Stents; Observational; All-Comers
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary artery stenting: All subjects who are candidates for coronary artery stenting, signed the Informed Consent Form and are eligible to receive a TAXUS Element stent will be evaluated for enrollment in this study.
  Interventions: Procedure: Coronary artery stenting

INTERVENTIONS:
Procedure: Coronary artery stenting — Coronary artery stenting with drug eluting stents
  Other Names: TAXUS Element

SUMMARY:
The goal of the TAXUS™ Element™ Paclitaxel-Eluting Coronary Stent System European Post-Approval Surveillance Study is to evaluate real world clinical outcomes data for the TAXUS™ Element™ Coronary Stent System in unselected patients in routine clinical practice.

DETAILED DESCRIPTION:
A prospective, open label, multi-center observational study with an all-comers enrollment approach of approximately 1000 subjects at up to 50 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

* According to Instructions For Use

Exclusion Criteria:

* Contraindications according to Instructions for Use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who are candidates for coronary artery stenting, signed the Informed Consent Form and are eligible to receive a TAXUS Element stent will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Target Vessel failure | 1 year
  Overall and TAXUS Element stent related Target Vessel Failure (TVF) rate (cardiac death, myocardial infarction (MI) related to target vessel and target vessel re-intervention (TVR)) at 12 months post stent implantation

SECONDARY OUTCOMES:
Stent Thrombosis | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Stent Thrombosis (ST) rate using Academic Research Consortium (ARC) definition (definite/probable with no censoring for Target Lesion Reintervention, (TLR)).
MACE | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Overall and TAXUS Element stent-related Major Adverse Cardiac Events (MACE) rates (cardiac death, MI, TVR).
Cardiac Death or MI | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Overall and TAXUS Element stent-related cardiac death or MI rates
TVR | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Overall and TAXUS Element stent-related TVR rates
Cardiac Death | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Overall and TAXUS Element stent-related cardiac death rates
MI | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Overall and TAXUS Element stent-related MI rates
All Death | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  All Death rates
Non-Cardiac Death | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  Non-Cardiac Death rates
All Death or MI | 30 days, 6 months, 12 months and then annually through 3 years post index stent implantation
  All Death or MI rates

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, Prof., Principal Investigator — Ospedale Ferrarotto, Via Citelli, 1, 95100 Catania, Italy; Peter Maurer, PhD, Study Director — Boston Scientific Corporation
Locations (37):
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - CHU de Charleroi - ISPPC, Charleroi
  - H-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- France (8):
  - CH Avignon, Avignon
  - CHU Besancon, Besançon
  - Centre Hospitalier Privé Saint Martin gds, Caen
  - CHU Grenoble, Grenoble
  - Hôpital Privé Clairval, Marseille
  - CHG de Pau, Pau
  - Clinique Saint-Hilaire Rouen, Rouen
  - Centre Hôpital Universitaire Rangueuil, Toulouse
- Germany (6):
  - Kardiocentrum Frankfurt, Frankfurt am Main, Hesse
  - Krankenhaus d. Barmherzigen Brüder, Trier, Rhineland-Palatinate
  - Klinikum Coburg gGmbH, Coburg
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Augusta Krankenhaus, Düsseldorf
  - Krankenhaus Landshut-Achdorf, Landshut
- Medical School of University PECS, Pécs, Hungary
- Galway University Hospital, Galway, Ireland
- Italy (4):
  - Ospedale Ferrarotto, Catania
  - Ospedale Cannizzaro, Catania
  - Ospedale Misericordia ASL 9, Grosseto
  - Azienda Ospedaliera Papardo, Messina
- P. Stradins University Hospital, Riga, Latvia
- Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki, Poland
- Spain (5):
  - Hospital General de Albacete, Albacete
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital General De Leon, León
  - Hospital La Paz, Madrid
  - H. Marques De Valdecilla, Santander
- United Kingdom (7):
  - Craigavon Hospital, Southern Trust, Craigavon, Northern Ireland
  - Royal Bournemouth General Hospital, Bournemouth
  - Lister, Hertfordshire
  - London Chest Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital NHS Trust, Norwich
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
Primary endpoint data presented at TCT 2014.

REFERENCES:
- [Result] Tamburino C, Capodanno D, Erglis A, Menown IB, Horvath IG, Moreno R, Gilbert TJ, Crowley JJ, Calabria P, Allocco DJ, Dawkins KD. One-year outcomes in unselected patients treated with a thin-strut, platinum-chromium, paclitaxel-eluting stent: primary endpoint results from the TAXUS Element European post-approval surveillance study (TE-PROVE). EuroIntervention. 2015 Mar;10(11):1261-6. doi: 10.4244/EIJY15M01_01. PMID 25572023